CLINICAL TRIAL: NCT02634307
Title: A Phase 3 Open Label Study to Evaluate the Long-term Safety and Tolerability of ALKS 8700 in Adults With Relapsing Remitting Multiple Sclerosis
Brief Title: A Study of ALKS 8700 in Adults With Relapsing Remitting Multiple Sclerosis (MS) EVOLVE-MS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK8700-A301; 2015-005160-41 (EudraCT Number)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: MS; Relapsing Remitting Multiple Sclerosis; RRMS; dimethyl fumarate; DMF
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALKS 8700 (Experimental): Oral capsules taken twice daily.
  Interventions: Drug: ALKS 8700

INTERVENTIONS:
Drug: ALKS 8700 — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of ALKS 8700 for the treatment of Relapsing Remitting Multiple Sclerosis (RRMS). The secondary objective of this study is to evaluate treatment effect over time in adult participants with RRMS treated with ALKS 8700.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a confirmed diagnosis of RRMS
* Neurologically stable with no evidence of relapse within 30 days prior to Visit 2

Exclusion Criteria:

* Subject is pregnant or breastfeeding or plans to become pregnant or begin breastfeeding at any point during the study and for 30 days after any study drug administration
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS
* History of clinically significant cardiovascular, pulmonary, gastrointestinal, dermatologic, psychiatric, neurologic (other than MS), and/or other major disease that would preclude participation in a clinical trial
* History of a myocardial infarction, including a silent myocardial infarction identified on ECG, or unstable angina

NOTE: Other protocol defined Includison/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1057 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (98):
- United States (64):
  - Alkermes Investigational Site, Cullman, Alabama
  - Alkermes Investigational Site, Phoenix, Arizona
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Berkeley, California
  - Alkermes Investigational Site, Loma Linda, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Basalt, Colorado
  - Alkermes Investigational Site, Centennial, Colorado
  - Alkermes Investigational Site, Denver, Colorado
  - Alkermes Investigational Site, Middlebury, Connecticut
  - Alkermes Investigational Site, Stamford, Connecticut
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Atlantis, Florida
  - Alkermes Investigational Site, Bradenton, Florida
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Naples, Florida
  - Alkermes Investigational Site, Ormond Beach, Florida
  - Alkermes Investigational Site, Sarasota, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Vero Beach, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Columbus, Georgia
  - Alkermes Investigational Site, Evanston, Illinois
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Des Moines, Iowa
  - Alkermes Investigational Site, Overland Park, Kansas
  - Alkermes Investigational Site, Lexington, Kentucky
  - Alkermes Investigational Site, Alexandria, Louisiana
  - Alkermes Investigational Site, Baton Rouge, Louisiana
  - Alkermes Investigational Site, Detroit, Michigan
  - Alkermes Investigational Site, Traverse City, Michigan
  - Alkermes Investigational Site, Golden Valley, Minnesota
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Albuquerque, New Mexico
  - Alkermes Investigational Site, Patchogue, New York
  - Alkermes Investigational Site, Plainview, New York
  - Alkermes Investigational Site, Stony Brook, New York
  - Alkermes Investigational Site, Syracuse, New York
  - Alkermes Investigational Site, Charlotte, North Carolina
  - Alkermes Investigational Site, Greensboro, North Carolina
  - Alkermes Investigational Site, Raleigh, North Carolina
  - Alkermes Investigational Site, Winston-Salem, North Carolina
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Columbus, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Medford, Oregon
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Greer, South Carolina
  - Alkermes Investigational Site, Rock Hill, South Carolina
  - Alkermes Investigational Site, Spartanburg, South Carolina
  - Alkermes Investigational Site, Cordova, Tennessee
  - Alkermes Investigational Site, Franklin, Tennessee
  - Alkermes Investigational Site, Knoxville, Tennessee
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Lubbock, Texas
  - Alkermes Investigational Site, Salt Lake City, Utah
  - Alkermes Investigational Site, Newport News, Virginia
  - Alkermes Investigational Site, Richmond, Virginia
  - Alkermes Investigational Site, Seattle, Washington
- Belgium (3):
  - Alkermes Investigational Site, Bruges
  - Alkermes Investigational Site, Fraiture
  - Alkermes Investigational Site, La Louvière
- Bulgaria (3):
  - Alkermes Investigational Site, Blagoevgrad
  - Alkermes Investigational Site, Pleven
  - Alkermes Investigational Site, Sofia
- Alkermes Investigational Site, Gatineau, Quebec, Canada
- Germany (5):
  - Alkermes Investigational Site, Berlin
  - Alkermes Investigational Site, Dresden
  - Alkermes Investigational Site, Leipzig
  - Alkermes Investigational Site, Ulm
  - Alkermes Investigational Site, Westerstede
- Poland (8):
  - Alkermes Investigational Site, Gdansk
  - Alkermes Investigational Site, Katowice
  - Alkermes Investigational Site, Kielce
  - Alkermes Investigational Site, Krakow
  - Alkermes Investigational Site, Lodz
  - Alkermes Investigational Site, Lublin
  - Alkermes Investigational Site, Plewiska
  - Alkermes Investigational Site, Szczecin
- Russia (2):
  - Alkermes Investigational Site, Krasnoyarsk
  - Alkermes Investigational Site, Nizhny Novgorod
- Serbia (3):
  - Alkermes Investigational Site, Belgrade
  - Alkermes Investigational Site, Kragujevac
  - Alkermes Investigational Site, Niš
- Spain (3):
  - Alkermes Investigational Site, Barcelona
  - Alkermes Investigational Site, Madrid
  - Alkermes Investigational Site, Santa Cruz de Tenerife
- Ukraine (6):
  - Alkermes Investigational Site, Dnipro
  - Alkermes Investigational Site, Ivano-Frankivsk
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Odesa
  - Alkermes Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Singer BA, Wray S, Gudesblatt M, Bumstead B, Ziemssen T, Bonnell A, Scaramozza M, Levin S, Shanmugasundaram M, Chen H, Mendoza JP, Lewin JB, Shankar SL. Lymphopenia is Not the Primary Therapeutic Mechanism of Diroximel Fumarate in Relapsing-Remitting Multiple Sclerosis: Subgroup Analyses of the EVOLVE-MS-1 Study. Neurol Ther. 2024 Aug;13(4):1273-1285. doi: 10.1007/s40120-024-00637-2. Epub 2024 Jun 27. PMID 38935202
- [Derived] Bowen JD, Stulc J, Hunter SF, Chen H, Lewin JB, Scaramozza M, Bozin I, Then Bergh F. Diroximel Fumarate in Patients with Relapsing-Remitting Multiple Sclerosis: NEDA-3 After Re-Baselining in the Phase 3 EVOLVE-MS-1 Study. Adv Ther. 2024 Aug;41(8):3396-3406. doi: 10.1007/s12325-024-02901-1. Epub 2024 Jun 15. PMID 38878121
- [Derived] Jiang T, Ziemssen T, Wray S, Shen C, Soderbarg K, Lewin JB, Bozin I, Freedman MS. Matching-Adjusted Indirect Comparisons of Diroximel Fumarate, Ponesimod, and Teriflunomide for Relapsing Multiple Sclerosis. CNS Drugs. 2023 May;37(5):441-452. doi: 10.1007/s40263-023-01002-x. Epub 2023 May 8. PMID 37155132
- [Derived] Wray S, Then Bergh F, Wundes A, Arnold DL, Drulovic J, Jasinska E, Bowen JD, Negroski D, Naismith RT, Hunter SF, Gudesblatt M, Chen H, Lyons J, Shankar SL, Kapadia S, Mendoza JP, Singer BA. Efficacy and Safety Outcomes with Diroximel Fumarate After Switching from Prior Therapies or Continuing on DRF: Results from the Phase 3 EVOLVE-MS-1 Study. Adv Ther. 2022 Apr;39(4):1810-1831. doi: 10.1007/s12325-022-02068-7. Epub 2022 Feb 24. PMID 35211872
- [Derived] Naismith RT, Wolinsky JS, Wundes A, LaGanke C, Arnold DL, Obradovic D, Freedman MS, Gudesblatt M, Ziemssen T, Kandinov B, Bidollari I, Lopez-Bresnahan M, Nangia N, Rezendes D, Yang L, Chen H, Liu S, Hanna J, Miller C, Leigh-Pemberton R. Diroximel fumarate (DRF) in patients with relapsing-remitting multiple sclerosis: Interim safety and efficacy results from the phase 3 EVOLVE-MS-1 study. Mult Scler. 2020 Nov;26(13):1729-1739. doi: 10.1177/1352458519881761. Epub 2019 Nov 4. PMID 31680631
- [Derived] Palte MJ, Wehr A, Tawa M, Perkin K, Leigh-Pemberton R, Hanna J, Miller C, Penner N. Improving the Gastrointestinal Tolerability of Fumaric Acid Esters: Early Findings on Gastrointestinal Events with Diroximel Fumarate in Patients with Relapsing-Remitting Multiple Sclerosis from the Phase 3, Open-Label EVOLVE-MS-1 Study. Adv Ther. 2019 Nov;36(11):3154-3165. doi: 10.1007/s12325-019-01085-3. Epub 2019 Sep 19. PMID 31538304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at investigational sites in North America and Europe from 10 December 2015 to 11 November 2021.
Pre-assignment Details: De Novo (who had not participated in any prior study of ALKS 8700) and Rollover participants (who had completed the Treatment Period of Study ALK8700-A302) were enrolled in this study.
Groups:
- De Novo: Participants who had not received ALKS 8700 or dimethyl fumarate (DMF) were administered ALKS 8700 231 milligrams (mg) capsules orally, twice daily (BID) on Days 1 to 7 followed by ALKS 8700 462 mg (as two 231 mg capsules) orally, BID from Day 8 up to Week 96.
- Rollover: ALKS 8700: Participants rolled over from study ALK870-A302 who had already received ALKS 8700 prior to Day 1 were administered ALKS 8700 462 mg (as two 231 mg capsules) orally, BID from Day 1 up to Week 96.
- Rollover: DMF: Participants rolled over from study ALK870-A302 who had already received DMF prior to Day 1 were administered ALKS 8700 462 mg (as two 231 mg capsules) orally, BID from Day 1 up to Week 96.
Period: Overall Study
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Started | 593 | 239 | 225
Safety Population | 593 | 239 | 225
Full Analysis Set (FAS) Population | 582 | 235 | 224
Completed | 468 | 168 | 164
Not Completed | 125 | 71 | 61
Not completed — Adverse Event | 50 | 24 | 14
Not completed — Lost to Follow-up | 21 | 5 | 6
Not completed — Pregnancy | 5 | 1 | 3
Not completed — Withdrawal by Subject | 38 | 24 | 18
Not completed — Non-Compliance with Study Drug | 0 | 2 | 2
Not completed — Lack of Efficacy | 1 | 5 | 3
Not completed — Physician Decision | 7 | 5 | 5
Not completed — Reason not Specified | 3 | 5 | 10

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Groups:
- De Novo: Participants who had not received ALKS 8700 or DMF were administered ALKS 8700 231 mg capsules orally, BID on Days 1 to 7 followed by ALKS 8700 462 mg (as two 231 mg capsules) orally, BID from Day 8 up to Week 96.
- Total: Total of all reporting groups
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF | Total
Number analyzed (Participants) | 593 | 239 | 225 | 1057
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.96) | 44.0 (11.00) | 43.7 (9.77) | 42.5 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 427 | 165 | 170 | 762
  Male | 166 | 74 | 55 | 295
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 5 | 10 | 40
  Not Hispanic or Latino | 568 | 234 | 215 | 1017
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 547 | 220 | 205 | 972
  Race: Black or African American | 37 | 19 | 16 | 72
  Race: Asian | 4 | 0 | 1 | 5
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Race: Other | 5 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAE is any AE that start or worsen on or after the date of first dose of study treatment. An SAE is any untoward medical occurrence that at any dose, results in death; in the view of the investigator places the participant at immediate risk of death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is a medically important event.
Time Frame: From first dose to two weeks after last dose of study drug (Up to 98 weeks)
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 593 | 239 | 225
Participants
  TEAEs | 519 | 212 | 207
  SAEs | 69 | 29 | 25

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Abnormalities
Description: Vital sign measurements included heart rate (low: <=50 beats per minute [bpm] and decrease >=15 bpm; High: >=120 bpm and increase >=15 bpm), systolic blood pressure (BP) (low: <=90 millimeters of mercury [mmHg] and decrease >=20 mmHg; High: >=180 mmHg and increase >=20 mmHg) and diastolic BP (low: <=50 mmHg and decrease >=15 mmHg; High: >=105 mmHg and increase >=15 mmHg).
Time Frame: From first dose to two weeks after last dose of study drug (Up to 98 weeks)
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700. 'Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure. 'Number Analyzed' signifies number of participants analyzed for the specified measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 582 | 238 | 225
Participants
  Systolic BP (Low: <=90 mmHg and decrease >=20 mmHg): number analyzed (Participants) | 581 | 237 | 224
  Systolic BP (Low: <=90 mmHg and decrease >=20 mmHg) | 15 | 4 | 2
  Systolic BP (High: >=180 mmHg and increase >=20 mmHg) | 3 | 2 | 1
  Diastolic BP (Low: <=50 mmHg and decrease >=15 mmHg): number analyzed (Participants) | 580 | 238 | 224
  Diastolic BP (Low: <=50 mmHg and decrease >=15 mmHg) | 10 | 2 | 4
  Diastolic BP (High: >=105 mmHg and increase >=15 mmHg): number analyzed (Participants) | 581 | 238 | 225
  Diastolic BP (High: >=105 mmHg and increase >=15 mmHg) | 6 | 2 | 2
  Heart Rate (Low: <=50 bpm and decrease >=15 bpm): number analyzed (Participants) | 579 | 235 | 225
  Heart Rate (Low: <=50 bpm and decrease >=15 bpm) | 5 | 1 | 2
  Heart Rate (High: >=120 bpm and increase >=15 bpm) | 1 | 1 | 2

3. Primary Outcome: Number of Participants With Potentially Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Potentially clinically significant QTcF values (>450 to <=480 millisecond [msec], >480 to <=500 msec) at any post-baseline visit during treatment period were reported.
Time Frame: From first dose to two weeks after last dose of study drug (Up to 98 weeks)
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700. 'Number of Participants Analyzed' signifies number of participants analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 576 | 237 | 223
Participants
  >450 - <=480 msec | 15 | 5 | 6
  >480 - <=500 msec | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Columbia Suicide Severity Rating Scale (C-SSRS) Score at Any Post-Baseline Visit
Description: The C-SSRS is a clinician-administered instrument that systematically assess suicidal ideation and behavior rating scale. It rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent). The scale identifies specific behaviors ranging from "preparatory acts or behavior" to "suicide" which may be indicative of an individual's intent to complete suicide.
Time Frame: Up to 98 weeks
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 593 | 239 | 225
Participants
  Suicidal Behavior: Preparatory acts or behavior | 0 | 0 | 0
  Suicidal Behavior: Aborted attempt | 0 | 0 | 0
  Suicidal Behavior: Interrupted attempt | 0 | 0 | 0
  Suicidal Behavior: Actual attempt | 1 | 0 | 0
  Suicidal Behavior: Completed suicide | 0 | 0 | 0
  Suicidal Ideation: Wish to be dead | 12 | 2 | 4
  Suicidal Ideation: Non-specific active suicidal thoughts | 8 | 2 | 2
  Suicidal Ideation: Active ideation without intention to act | 2 | 0 | 1
  Suicidal Ideation: Active ideation with some intent to act without a plan | 1 | 0 | 0
  Suicidal Ideation: Active ideation with a specific plan and intent | 1 | 0 | 0
  Non-Suicidal Self-Injurious Behavior | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities
Description: Laboratory assessments included hematology, biochemistry, and urinalysis. Abnormality criteria: >=3xupper limit of normal (ULN) in alanine aminotransferase, aspartate aminotransferase; In millimoles per liter (mmol/L) [bicarbonate<15/>31, chloride<=90, potassium<3/>5.5, sodium<130/>150]; In mg per decilitre(mg/dL) {total bilirubin>=2.0, calcium<8.2/>12, total cholesterol>300, creatinine>=2.0, glucose<50/>200, cholesterol: High density lipoprotein (HDL)<=30, low density lipoprotein (LDL)>=160, triglycerides>=120 [female(F)]/>=160 [male(M)], urate>9/>8(F), blood urea nitrogen>30}; >3xULN in creatine kinase, lactate dehydrogenase; Hematocrit <=32(F)/<=37(M) percentage(%),3 point decrease from baseline; Hemoglobin<=9.5(F)/<=11.5(M)g/dL; Lymphocytes<0.5x10^9/L; In 10^3/microliter(uL) [Eosinophils>1; Absolute neutrophils<1.5; Platelets<75.1/>=700; Leukocytes<=2.8/>=16]; Albumin/creatinine>200g/kilograms(kg); Beta-2 microglobulin >0.3milligrams/liter(mg/L); Glucose/protein at least 2+.
Time Frame: From first dose to two weeks after last dose of study drug (Up to 98 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 582 | 238 | 225
Participants
  Alanine Aminotransferase (U/L) >=3 x ULN: number analyzed (Participants) | 581 | 237 | 223
  Alanine Aminotransferase (U/L) >=3 x ULN | 13 | 6 | 1
  Aspartate Aminotransferase (U/L) >=3 x ULN: number analyzed (Participants) | 581 | 237 | 223
  Aspartate Aminotransferase (U/L) >=3 x ULN | 8 | 3 | 1
  Bicarbonate <15 mmol/L: number analyzed (Participants) | 582 | 237 | 225
  Bicarbonate <15 mmol/L | 3 | 0 | 0
  Bicarbonate >31 mmol/L: number analyzed (Participants) | 582 | 237 | 224
  Bicarbonate >31 mmol/L | 13 | 1 | 3
  Bilirubin, Total >=2.0 mg/dL: number analyzed (Participants) | 582 | 238 | 224
  Bilirubin, Total >=2.0 mg/dL | 2 | 1 | 0
  Calcium <8.2 mg/dL: number analyzed (Participants) | 580 | 238 | 225
  Calcium <8.2 mg/dL | 2 | 0 | 0
  Calcium >12 mg/dL | 0 | 1 | 0
  Cholesterol, Total >300 mg/dL: number analyzed (Participants) | 574 | 237 | 223
  Cholesterol, Total >300 mg/dL | 23 | 8 | 8
  Creatine Kinase (U/L) >3 x ULN: number analyzed (Participants) | 582 | 235 | 224
  Creatine Kinase (U/L) >3 x ULN | 26 | 11 | 8
  Chloride <=90 mmol/L: number analyzed (Participants) | 582 | 237 | 225
  Chloride <=90 mmol/L | 1 | 0 | 0
  Creatinine >=2.0 mg/dL: number analyzed (Participants) | 581 | 238 | 225
  Creatinine >=2.0 mg/dL | 1 | 0 | 2
  Glucose <50 mg/dL: number analyzed (Participants) | 579 | 237 | 225
  Glucose <50 mg/dL | 4 | 6 | 4
  Glucose >200 mg/dL: number analyzed (Participants) | 581 | 237 | 224
  Glucose >200 mg/dL | 6 | 5 | 4
  HDL Cholesterol <=30 mg/dL: number analyzed (Participants) | 575 | 238 | 221
  HDL Cholesterol <=30 mg/dL | 13 | 6 | 3
  Potassium <3 mmol/L | 1 | 0 | 0
  Potassium >5.5 mmol/L: number analyzed (Participants) | 577 | 237 | 225
  Potassium >5.5 mmol/L | 39 | 8 | 16
  Lactate Dehydrogenase (U/L) >3 x ULN: number analyzed (Participants) | 579 | 238 | 225
  Lactate Dehydrogenase (U/L) >3 x ULN | 1 | 0 | 0
  LDL Cholesterol >=160 mg/dL: number analyzed (Participants) | 521 | 226 | 207
  LDL Cholesterol >=160 mg/dL | 69 | 27 | 29
  Sodium <130 mmol/L: number analyzed (Participants) | 581 | 238 | 225
  Sodium <130 mmol/L | 1 | 0 | 0
  Sodium >150 mmol/L | 3 | 0 | 0
  Triglycerides >=120 mg/dL (Female): number analyzed (Participants) | 270 | 102 | 111
  Triglycerides >=120 mg/dL (Female) | 123 | 45 | 61
  Triglycerides >=160 mg/dL (Male): number analyzed (Participants) | 116 | 60 | 41
  Triglycerides >=160 mg/dL (Male) | 54 | 32 | 24
  Urate >9 mg/dL: number analyzed (Participants) | 580 | 236 | 225
  Urate >9 mg/dL | 10 | 5 | 2
  Urate >8 mg/dL (Female): number analyzed (Participants) | 415 | 164 | 168
  Urate >8 mg/dL (Female) | 8 | 3 | 4
  Blood Urea Nitrogen >30 mg/dL: number analyzed (Participants) | 582 | 237 | 225
  Blood Urea Nitrogen >30 mg/dL | 5 | 3 | 2
  Eosinophils >1x10^3/uL: number analyzed (Participants) | 581 | 236 | 211
  Eosinophils >1x10^3/uL | 8 | 3 | 1
  Hematocrit <=32% and 3 point decrease from baseline (Female): number analyzed (Participants) | 410 | 160 | 165
  Hematocrit <=32% and 3 point decrease from baseline (Female) | 18 | 5 | 8
  Hematocrit <=37% and 3 point decrease from baseline (Male): number analyzed (Participants) | 163 | 72 | 53
  Hematocrit <=37% and 3 point decrease from baseline (Male) | 6 | 4 | 3
  Hemoglobin <=9.5 g/dL (Female): number analyzed (Participants) | 414 | 164 | 169
  Hemoglobin <=9.5 g/dL (Female) | 5 | 1 | 3
  Hemoglobin <=11.5 g/dL (Male): number analyzed (Participants) | 164 | 72 | 55
  Hemoglobin <=11.5 g/dL (Male) | 2 | 1 | 0
  Lymphocytes <0.5x10^9/L | 47 | 25 | 24
  Neutrophils, Absolute <1.5x10^3/uL: number analyzed (Participants) | 580 | 236 | 224
  Neutrophils, Absolute <1.5x10^3/uL | 39 | 10 | 13
  Platelets <75.1x10^3/uL: number analyzed (Participants) | 581 | 238 | 225
  Platelets <75.1x10^3/uL | 2 | 0 | 1
  Platelets >=700x10^3/uL: number analyzed (Participants) | 581 | 238 | 225
  Platelets >=700x10^3/uL | 0 | 0 | 0
  Leukocytes <=2.8x10^3/uL: number analyzed (Participants) | 581 | 238 | 225
  Leukocytes <=2.8x10^3/uL | 45 | 17 | 15
  Leukocytes >=16x10^3/uL: number analyzed (Participants) | 581 | 238 | 224
  Leukocytes >=16x10^3/uL | 4 | 5 | 5
  Albumin/Creatinine >200 g/kg: number analyzed (Participants) | 581 | 237 | 225
  Albumin/Creatinine >200 g/kg | 15 | 8 | 5
  Beta-2 Microglobulin >0.300 mg/L: number analyzed (Participants) | 568 | 228 | 214
  Beta-2 Microglobulin >0.300 mg/L | 95 | 32 | 31
  Glucose at least 2+: number analyzed (Participants) | 579 | 237 | 223
  Glucose at least 2+ | 10 | 4 | 3
  Protein at least 2+: number analyzed (Participants) | 581 | 238 | 223
  Protein at least 2+ | 15 | 4 | 9

6. Other Pre Specified Outcome: Annualized Relapse Rate (ARR)
Description: Relapse was defined as new or recurrent neurologic symptoms, not associated with fever or infection, lasting for at least 24 hours, accompanied by one or more of the following: New objective neurological findings upon examination by the treating neurologist that are functionally consistent with findings on the Expanded Disability Status Scale [EDSS] (performed within 7 days of onset of symptoms) with an increase over the prior visit of ≥ 0.5 for the total score, an increase of ≥ 2 in 1 functional system (FS), except bladder/cognitive changes, and/or, an increase of ≥ 1 in 2 FS, except bladder/cognitive changes. The relapse rate for an individual participant was calculated as the number of relapses for that participant divided by the number of participant-years followed. The ARR for each enrollment group was calculated as the total number of relapses experienced in the group divided by the total number of participant-years on study.
Time Frame: Up to 96 weeks
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Measure: Number; unit: relapses per participant year
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 593 | 239 | 225
relapses per participant year | 0.14 | 0.11 | 0.13

7. Other Pre Specified Outcome: Percentage of Participants With Multiple Sclerosis (MS) Relapse
Description: Relapse was defined as new or recurrent neurologic symptoms, not associated with fever or infection, lasting for at least 24 hours, accompanied by one or more of the following: New objective neurological findings upon examination by the treating neurologist that are functionally consistent with findings on the EDSS (performed within 7 days of onset of symptoms) with an increase over the prior visit of ≥ 0.5 for the total score, an increase of ≥ 2 in 1 FS, except bladder/cognitive changes, and/or, an increase of ≥ 1 in 2 FS, except bladder/cognitive changes.
Time Frame: Up to 96 weeks
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Measure: Number; unit: percentage of participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 593 | 239 | 225
percentage of participants | 17.66 | 16.66 | 18.30

8. Other Pre Specified Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score
Description: The EDSS is used to measure and evaluate MS participants' level of functioning. The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic examination; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to MS. Higher scores indicate more disability. Positive change from baseline indicates more disability.
Time Frame: Baseline up to Week 96
Population: FAS included all participants who received at least one dose of ALKS 8700 and had at least one post-baseline efficacy assessment. 'Number Analyzed' signifies number of participants analyzed for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 582 | 235 | 224
score on a scale
  Baseline | 2.71 (1.457) | 2.64 (1.481) | 2.71 (1.445)
  Change From Baseline at Week 12: number analyzed (Participants) | 576 | 232 | 224
  Change From Baseline at Week 12 | -0.01 (0.490) | -0.03 (0.548) | 0.05 (0.557)
  Change From Baseline at Week 24: number analyzed (Participants) | 549 | 217 | 214
  Change From Baseline at Week 24 | 0.00 (0.518) | -0.02 (0.603) | -0.01 (0.696)
  Change From Baseline at Week 36: number analyzed (Participants) | 531 | 212 | 209
  Change From Baseline at Week 36 | 0.01 (0.558) | -0.01 (0.597) | -0.03 (0.733)
  Change From Baseline at Week 48: number analyzed (Participants) | 521 | 203 | 202
  Change From Baseline at Week 48 | 0.03 (0.614) | -0.01 (0.579) | 0.00 (0.702)
  Change From Baseline at Week 60: number analyzed (Participants) | 511 | 192 | 190
  Change From Baseline at Week 60 | 0.04 (0.617) | -0.02 (0.643) | -0.02 (0.633)
  Change From Baseline at Week 72: number analyzed (Participants) | 498 | 189 | 184
  Change From Baseline at Week 72 | 0.05 (0.617) | -0.04 (0.639) | 0.08 (0.713)
  Change From Baseline at Week 84: number analyzed (Participants) | 486 | 174 | 177
  Change From Baseline at Week 84 | 0.07 (0.641) | -0.03 (0.616) | -0.02 (0.759)
  Change From Baseline at Week 96: number analyzed (Participants) | 478 | 172 | 166
  Change From Baseline at Week 96 | 0.07 (0.631) | -0.01 (0.775) | 0.03 (0.735)

9. Other Pre Specified Outcome: Change From Baseline in Timed 25-Foot Walk Test (T25-FW) Score
Description: The T25-FW is a reliable quantitative mobility and leg function performance test based on a timed 25-foot walk. The participant was directed to one end of a clearly marked 25-foot course and was instructed to walk 25 feet as quickly as possible, but safely. Participants were allowed to use assistive devices (canes, crutches, walkers) as needed. The time was calculated from when the lead foot crosses the start point to when the participant had reached the 25-foot mark. The task was immediately administered again by having the participant walk back the same distance. The score for the T25-FW was calculated as the average of the 2 completed trials. A negative change from Baseline indicates improvement.
Time Frame: Baseline up to Week 96
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 582 | 235 | 224
seconds
  Baseline | 5.875 [4.900 to 7.500] | 5.350 [4.500 to 6.850] | 5.635 [4.575 to 7.020]
  Change From Baseline at Week 12: number analyzed (Participants) | 579 | 232 | 224
  Change From Baseline at Week 12 | -0.050 [-0.450 to 0.250] | 0.000 [-0.250 to 0.350] | 0.000 [-0.425 to 0.375]
  Change From Baseline at Week 24: number analyzed (Participants) | 551 | 218 | 214
  Change From Baseline at Week 24 | 0.000 [-0.450 to 0.300] | -0.050 [-0.350 to 0.400] | 0.000 [-0.450 to 0.400]
  Change From Baseline at Week 36: number analyzed (Participants) | 526 | 213 | 209
  Change From Baseline at Week 36 | -0.050 [-0.500 to 0.300] | -0.100 [-0.450 to 0.350] | 0.000 [-0.500 to 0.500]
  Change From Baseline at Week 48: number analyzed (Participants) | 517 | 199 | 201
  Change From Baseline at Week 48 | 0.000 [-0.450 to 0.400] | 0.000 [-0.450 to 0.350] | -0.050 [-0.450 to 0.550]
  Change From Baseline at Week 60: number analyzed (Participants) | 511 | 194 | 191
  Change From Baseline at Week 60 | -0.050 [-0.600 to 0.400] | -0.090 [-0.550 to 0.300] | 0.000 [-0.550 to 0.550]
  Change From Baseline at Week 72: number analyzed (Participants) | 499 | 185 | 183
  Change From Baseline at Week 72 | 0.000 [-0.550 to 0.500] | -0.050 [-0.600 to 0.350] | 0.000 [-0.550 to 0.600]
  Change From Baseline at Week 84: number analyzed (Participants) | 486 | 174 | 173
  Change From Baseline at Week 84 | -0.050 [-0.600 to 0.450] | -0.075 [-0.500 to 0.300] | 0.000 [-0.500 to 0.700]
  Change From Baseline at Week 96: number analyzed (Participants) | 476 | 169 | 165
  Change From Baseline at Week 96 | -0.050 [-0.550 to 0.400] | -0.050 [-0.500 to 0.400] | 0.000 [-0.450 to 0.650]

10. Other Pre Specified Outcome: Change From Baseline in the EuroQol 5-Dimension 5-Level Visual Analog Scale (EQ-5D-5L VAS) Score
Description: The EQ-5D-5L is an instrument designed to assess decrements in health. The EQ-5D-5L includes a VAS and a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response categories corresponding to the level of severity (i.e., no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems). The EQ-5D-5L VAS records the participant's self-rated health on a vertical visual analogue scale numbered from 100 (best health imagined) to 0 (worst health imagined). Higher scores indicate good health. Positive change from baseline indicates improved health.
Time Frame: Baseline up to Week 96
Population: FAS included all participants who received at least one dose of ALKS 8700 and had at least one post-baseline efficacy assessment. 'Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure. 'Number Analyzed' signifies number of participants analyzed for this outcome measure at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 581 | 232 | 221
score on a scale
  Baseline | 73.7 (17.48) | 80.3 (14.65) | 80.0 (16.26)
  Change From Baseline at Week 24: number analyzed (Participants) | 560 | 222 | 216
  Change From Baseline at Week 24 | 1.0 (15.30) | -1.6 (12.24) | -1.6 (12.31)
  Change From Baseline at Week 48: number analyzed (Participants) | 523 | 204 | 202
  Change From Baseline at Week 48 | 0.3 (15.27) | -2.8 (10.68) | -1.9 (12.48)
  Change From Baseline at Week 72: number analyzed (Participants) | 498 | 192 | 187
  Change From Baseline at Week 72 | 1.3 (14.85) | -2.8 (11.97) | -2.1 (12.50)
  Change From Baseline at Week 96: number analyzed (Participants) | 481 | 173 | 169
  Change From Baseline at Week 96 | 0.6 (14.59) | -4.2 (12.35) | -3.7 (14.71)

11. Other Pre Specified Outcome: Change From Baseline in the EQ-5D-5L Index Score
Description: The EQ-5D-5L is an instrument designed to assess decrements in health. The EQ-5D-5L includes a VAS and a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response categories corresponding to the level of severity (i.e., no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems). The 5-item index score is transformed into a utility score between 0 (worst health state) and 1 (best health state). Higher scores indicate good health. Positive change from baseline indicates improved health.
Time Frame: Baseline up to Week 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 581 | 232 | 221
score on a scale
  Baseline | 0.793 (0.137) | 0.841 (0.128) | 0.837 (0.128)
  Change From Baseline at Week 24: number analyzed (Participants) | 560 | 222 | 216
  Change From Baseline at Week 24 | -0.002 (0.110) | -0.018 (0.085) | -0.035 (0.096)
  Change From Baseline at Week 48: number analyzed (Participants) | 522 | 203 | 202
  Change From Baseline at Week 48 | -0.006 (0.108) | -0.026 (0.086) | -0.037 (0.101)
  Change From Baseline at Week 72: number analyzed (Participants) | 498 | 192 | 187
  Change From Baseline at Week 72 | -0.010 (0.109) | -0.030 (0.108) | -0.036 (0.110)
  Change From Baseline at Week 96: number analyzed (Participants) | 481 | 173 | 168
  Change From Baseline at Week 96 | -0.009 (0.114) | -0.042 (0.109) | -0.057 (0.117)

12. Other Pre Specified Outcome: Change From Baseline in the 12-item Short Form Health Survey (SF-12) Score
Description: The SF-12 uses 12 questions to measure functional health and well-being from the study participant's perspective across eight domains: physical functioning, role, bodily pain, general health perceptions, vitality, social functioning, emotional role, and mental health. Mental and physical composite scores (MCS & PCS) are computed using the scores of twelve questions and range from 0 to 100, where a higher score indicates better health. Positive change from baseline indicates improved health.
Time Frame: Baseline up to Week 96
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 582 | 235 | 224
score on a scale
  PCS: Baseline: number analyzed (Participants) | 578 | 235 | 224
  PCS: Baseline | 42.90 (10.662) | 44.68 (10.629) | 45.03 (10.720)
  PCS: Change From Baseline at Week 24: number analyzed (Participants) | 555 | 221 | 216
  PCS: Change From Baseline at Week 24 | 0.35 (7.329) | -0.28 (6.893) | -1.00 (6.248)
  PCS: Change From Baseline at Week 48: number analyzed (Participants) | 523 | 203 | 200
  PCS: Change From Baseline at Week 48 | 0.22 (6.804) | -0.04 (7.428) | -1.62 (6.546)
  PCS: Change From Baseline at Week 72: number analyzed (Participants) | 491 | 192 | 185
  PCS: Change From Baseline at Week 72 | 0.04 (7.341) | -0.27 (7.902) | -1.25 (6.849)
  PCS: Change From Baseline at Week 96: number analyzed (Participants) | 476 | 173 | 169
  PCS: Change From Baseline at Week 96 | 0.48 (7.154) | -0.28 (7.095) | -1.44 (7.191)
  MCS: Baseline: number analyzed (Participants) | 578 | 235 | 224
  MCS: Baseline | 47.75 (10.345) | 50.90 (8.926) | 51.14 (9.299)
  MCS: Change From Baseline at Week 24: number analyzed (Participants) | 555 | 221 | 216
  MCS: Change From Baseline at Week 24 | 0.29 (8.745) | -2.12 (7.962) | -1.69 (8.415)
  MCS: Change From Baseline at Week 48: number analyzed (Participants) | 523 | 203 | 200
  MCS: Change From Baseline at Week 48 | -0.62 (9.412) | -2.57 (8.059) | -2.20 (9.386)
  MCS: Change From Baseline at Week 72: number analyzed (Participants) | 491 | 192 | 185
  MCS: Change From Baseline at Week 72 | -0.34 (9.866) | -2.63 (7.786) | -3.50 (9.663)
  MCS: Change From Baseline at Week 96: number analyzed (Participants) | 476 | 173 | 169
  MCS: Change From Baseline at Week 96 | -0.35 (9.517) | -2.93 (8.681) | -3.57 (10.582)

13. Other Pre Specified Outcome: Time to Onset of 12-week Confirmed Disability Progression
Description: The time to onset of 12-week confirmed disability progression is defined as the time from baseline to the first disability progression that is confirmed at the next regularly scheduled visit ≥ 12 weeks after the initial disability progression. Disability progression is defined by one of the following: an EDSS increase of at least 1.5 points from baseline EDSS = 0, an EDSS increase of at least a 1.0 point from baseline EDSS between 1.0 and 5.5 (inclusive), or an EDSS increase of at least 0.5 points from baseline EDSS = 6.0.
Time Frame: Up to Week 96
Population: FAS included all participants who received at least one dose of ALKS 8700 and had at least one post-baseline efficacy assessment. 'Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 47 | 22 | 23
days | 250.0 [91.0 to 420.0] | 254.5 [89.0 to 419.0] | 176.0 [89.0 to 333.0]

14. Other Pre Specified Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA) at Week 96
Description: The definition of NEDA-3 encompasses a combination of the following 3 related measures of disease activity: No relapses, no confirmed disability progression sustained for 12 weeks as measured on EDSS, and no magnetic resonance imaging (MRI) disease activity, defined as no gadolinium-enhancing (GdE) lesions and no new or enlarging T2 lesions. The definition of NEDA-4 was the above definition of NEDA-3 with the addition of a mean annualized rate of brain volume loss of less than 0.4% where annualized rate of brain volume loss was derived from percentage brain volume change (PBVC) from baseline and was calculated as ([PBVC/100+1]^[365.25/days]-1) × 100.
Time Frame: Week 96
Population: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700. 'Number Analyzed' signifies number of participants analyzed for this outcome measure at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
Number analyzed (Participants) | 487 | 185 | 185
percentage of participants
  NEDA-3 | 24.8 | 34.6 | 28.6
  NEDA-4: number analyzed (Participants) | 419 | 158 | 160
  NEDA-4 | 14.3 | 15.2 | 11.9

ADVERSE EVENTS:
Time Frame: From first dose to two weeks after last dose of study drug (Up to 98 weeks)
Description: Safety Analysis Set included all enrolled participants who received at least one dose of ALKS 8700.
Arm/Group | De Novo | Rollover: ALKS 8700 | Rollover: DMF
All-Cause Mortality (participants affected / at risk) | 3/593 | 1/239 | 0/225
Serious Adverse Events (participants affected / at risk) | 69/593 | 29/239 | 25/225
Other Adverse Events (participants affected / at risk) | 461/593 | 186/239 | 189/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=593) | Rollover: ALKS 8700 (N=239) | Rollover: DMF (N=225)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestatic liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
VIIIth nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cerebellar embolism (Nervous system disorders) | 0 | 0 | 1
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 32 | 19 | 10
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Uhthoff's phenomenon (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo (N=593) | Rollover: ALKS 8700 (N=239) | Rollover: DMF (N=225)
Lymphopenia (Blood and lymphatic system disorders) | 51 | 35 | 38
Abdominal pain upper (Gastrointestinal disorders) | 30 | 5 | 5
Constipation (Gastrointestinal disorders) | 26 | 10 | 13
Diarrhoea (Gastrointestinal disorders) | 66 | 18 | 25
Nausea (Gastrointestinal disorders) | 45 | 12 | 15
Fatigue (General disorders) | 39 | 26 | 22
Nasopharyngitis (Infections and infestations) | 86 | 24 | 27
Sinusitis (Infections and infestations) | 34 | 17 | 14
Upper respiratory tract infection (Infections and infestations) | 76 | 42 | 35
Urinary tract infection (Infections and infestations) | 55 | 25 | 24
Alanine aminotransferase increased (Investigations) | 30 | 17 | 11
Lymphocyte count decreased (Investigations) | 21 | 13 | 12
Urine albumin/creatinine ratio increased (Investigations) | 13 | 6 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 18 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 18 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 | 11 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 12 | 12
Dizziness (Nervous system disorders) | 31 | 12 | 14
Headache (Nervous system disorders) | 49 | 23 | 24
Hypoaesthesia (Nervous system disorders) | 19 | 13 | 11
Multiple sclerosis relapse (Nervous system disorders) | 93 | 47 | 44
Depression (Psychiatric disorders) | 23 | 14 | 13
Erythema (Skin and subcutaneous tissue disorders) | 38 | 8 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 52 | 8 | 10
Flushing (Vascular disorders) | 226 | 33 | 29
Hypertension (Vascular disorders) | 13 | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT02634307/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT02634307/SAP_001.pdf